CLINICAL TRIAL: NCT04305912
Title: Comparison of Verofilcon A Daily Disposable Lenses to Somofilcon A Daily Disposable Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: EX-MKTG-113
Record Dates: First submitted 2020-03-09; First posted 2020-03-12 (Actual); Results first posted 2022-02-11 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-02

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- somofilcon A (Experimental): Subjects will be randomized to wear somofilcon A daily disposable lenses for one week and then switch to verofilcon A daily disposable lenses for one week.
  Interventions: Device: somofilcon A
- verofilcon A (Active Comparator): Subjects will be randomized to wear verofilcon A daily disposable lenses for one week and then switch to somofilcon A daily disposable lenses for one week.
  Interventions: Device: verofilcon A

INTERVENTIONS:
Device: somofilcon A — Subjects will be randomized to wear somofilcon A daily disposable lenses.
  Other Names: Clariti 1 Day
  Arms: somofilcon A
Device: verofilcon A — Subjects will be randomized to wear verofilcon A daily disposable lenses.
  Other Names: Precision 1
  Arms: verofilcon A

SUMMARY:
The objective of the study is to evaluate and compare the performance of verofilcon A to somofilcon A when worn on a daily disposable modality over a period of approximately one week each.

DETAILED DESCRIPTION:
The study is a prospective, double masked (investigator and participant), bilateral, randomized,one week cross-over dispensing study, which evaluates somofilcon A (test lens) and verofilcon A (control lens).

ELIGIBILITY:
Inclusion Criteria:

-

A person is eligible for inclusion in the study if he/she:

1. Is at least 17 years of age and has full legal capacity to volunteer;
2. Has read and signed an information consent letter;
3. Is willing and able to follow instructions and maintain the appointment schedule;
4. Habitually wears soft contact lenses in daily wear, for minimum of 6-months;
5. Is correctable to a visual acuity of 20/40 or better (in each eye) with the study lenses;
6. Has an astigmatism of ≤ 1.00 D in subjective refraction;
7. Can be fit with study contact lenses with a power between -2.00 and -5.00 DS;
8. Demonstrates an acceptable fit with the study lenses;
9. Habitually wears single vision soft contact lenses for at least 8 hours per day, 5 days a week, and is willing to wear contact lenses for at least 12 hours a day in the study.

Exclusion Criteria:

-

A person may be excluded from the study if he/she:

1. Is participating in any concurrent clinical or research study;
2. Has any known active* ocular disease and/or infection;
3. Has a systemic condition that in the opinion of the investigator may affect a study outcome variable;
4. Is using any systemic or topical medications that in the opinion of the investigator may affect a study outcome variable;
5. Has known sensitivity to the diagnostic pharmaceuticals to be used in the study;
6. Is pregnant, lactating or planning a pregnancy at the time of enrolment because the associated hormonal changes cause changes in the tear layer which impact contact lens comfort. Verbal confirmation at the screening visit is sufficient;
7. Is aphakic;
8. Has undergone refractive error surgery;
9. Is an employee of the Centre for Ocular Research & Education;
10. Has participated in the BOXER (i.e. EX-MKTG-107, phases 1 or 2) or MIKI (EX-MKTG-114) Study;
11. Has participated in any clinical trials within a week prior to the study.

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2020-02-19 (Actual); Primary Completion 2021-08-28 (Actual); Study Completion 2021-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lyndon Jones, PhD FCOptom, Principal Investigator — University of Waterloo
Locations (1):
- University of Waterloo, Waterloo, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Somofilcon A Then Verofilcon A: Subjects will be randomized to wear somofilcon A daily disposable lenses for one week and then switch to verofilcon A daily disposable lenses for one week.
- Verofilcon A the Somofilcon A: Subjects will be randomized to wear verofilcon A daily disposable lenses for one week and then switch to somofilcon A daily disposable lenses for one week.
Period: First Intervention
Arm/Group | Somofilcon A Then Verofilcon A | Verofilcon A the Somofilcon A
Started | 26 | 25
Completed | 24 | 24
Not Completed | 2 | 1
Not completed — COVID-19 Suspension | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1
Period: Second Intervention
Arm/Group | Somofilcon A Then Verofilcon A | Verofilcon A the Somofilcon A
Started | 24 | 24
Completed | 24 | 23
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: Subjects will be randomized to wear somofilcon A daily disposable lenses and verofilcon A daily disposable lenses for one week.
Arm/Group | Overall Study
Number analyzed (Participants) | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 50
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.8 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 51

OUTCOME MEASURES:

1. Primary Outcome: Subjective Ratings for Lens Handling for Lens Insertion
Description: Subjective ratings for Lens handling for lens insertion (0 - 10 integer scale), (0- very difficult, 10- very easy).
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Somofilcon A: Subjects will be randomized to wear somofilcon A daily disposable lenses for one week.
- Verofilcon A: Subjects will be randomized to wear verofilcon A daily disposable lenses for one week.
Arm/Group | Somofilcon A | Verofilcon A
Number analyzed (Participants) | 47 | 47
units on a scale | 9.3 (0.9) | 9.2 (1.2)

2. Primary Outcome: Subjective Ratings for Lens Handling for Lens Removal
Description: Subjective ratings for Lens handling for lens removal (0 - 10 integer scale), (0-very difficult, 10- very easy).
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Somofilcon A | Verofilcon A
Number analyzed (Participants) | 47 | 47
units on a scale | 9.1 (1.3) | 8.8 (1.9)

3. Secondary Outcome: Lens Fit - Centration
Description: Lens Fit Centration was measured on a scale of 0-3 (0-optimal, 1-slight decentration, 2-moderate decentration but not encroaching limbus, 3- excessive & occasionally encroaching limbus)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Somofilcon A | Verofilcon A
Number analyzed (Participants) | 47 | 47
units on a scale | 0.7 (0.7) | 0.4 (0.5)

4. Secondary Outcome: Lens Fit - Centration
Description: as for outcome 3
Time Frame: 1-week
Population: One subject missed follow-up assessment for lens-fit centration.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Somofilcon A | Verofilcon A
Number analyzed (Participants) | 46 | 46
units on a scale | 0.5 (0.6) | 0.3 (0.5)

5. Secondary Outcome: Lens Fit - Post-blink Movement
Description: Post-blink lens movement was measured using an eyepiece reticule while viewing the contact lens in vivo at 8x magnification in primary gaze, in 0.1mm steps
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Somofilcon A | Verofilcon A
Number analyzed (Participants) | 47 | 47
mm | 0.2 (0.1) | 0.2 (0.1)

6. Secondary Outcome: Lens Fit - Post-blink Movement
Description: as for outcome 5
Time Frame: 1-week
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Somofilcon A | Verofilcon A
Number analyzed (Participants) | 47 | 47
mm | 0.2 (0.1) | 0.2 (0.1)

7. Secondary Outcome: Lens Fit - Lens Push-up Tightness
Description: The lens push-up tightness was graded using a 0 - 100 scale (5% steps) where 0% = falls from cornea without lid support, 50% = optimum and 100% = no movement
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Somofilcon A | Verofilcon A
Number analyzed (Participants) | 47 | 47
units on a scale | 50 (4) | 49 (5)

8. Secondary Outcome: Lens Fit - Lens Push-up Tightness
Description: as for outcome 7
Time Frame: 1-week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Somofilcon A | Verofilcon A
Number analyzed (Participants) | 47 | 47
units on a scale | 51 (5) | 51 (5)

ADVERSE EVENTS:
Time Frame: From dispense to 1 week on each lens, a total of two weeks.
Arm/Group | Somofilcon A | Verofilcon A
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/51
Other Adverse Events (participants affected / at risk) | 2/51 | 1/51
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Somofilcon A (N=51) | Verofilcon A (N=51)
Conjunctival Hyperemia (Eye disorders) | 1 (1) | 0 (0)
Mild Ocular Redness (Eye disorders) | 1 (1) | 0 (0)
Headache (Eye disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-16): https://cdn.clinicaltrials.gov/large-docs/12/NCT04305912/Prot_SAP_000.pdf